CLINICAL TRIAL: NCT06264479
Title: Prospective Evaluation of AI R&D Tool for Patient Stratification: a Trial for Renal Immuno-oncology Model Experimental Evaluation 2
Acronym: PEAR-TREE2
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Ourotech, Inc. (Industry)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other); Cambridge University Hospitals NHS Trust (Unknown); East & North Herts NHS Trust (Unknown); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PEAR-TREE2
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Kidney Cancer; Renal Cell Cancer Metastatic
Keywords: computer vision; cell culture; microtumor; functional testing; predictive biomarker; immuno-oncology
MeSH Terms: conditions — Kidney Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor cores and blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial Cohort: Patients with advanced or metastatic kidney cancer, due to start a new line of systemic therapy (targeted drug, immunotherapy, etc.)
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Patients undergo a biopsy from a lesion, and give 40ml of blood

SUMMARY:
Pear Bio has developed a predictive biomarker technology that combines 3D cell culture, microscopy and computer vision to measure the response of an individual patient's tumor sample to different systemic therapy regimens that are tested simultaneously ex vivo.

This study will recruit patients with advanced or metastatic kidney cancer who are due to start a clinically-indicated new line of therapy.

The oncologist will be blinded to the response on the Pear Bio test (the test will be run in parallel with the patient's treatment). The primary objective of this study is to establish the sensitivity and specificity of Pear Bio's test results against patient outcomes (objective response, progression-free survival, depth and duration of response, overall survival).

DETAILED DESCRIPTION:
This is a multicenter, international, observational pilot study that aims to determine the accuracy of a new assay, the Pear Bio test, in predicting response rate (ORR) in patients receiving standard of care systemic therapies for kidney cancer. Patients will undergo an additional, mandatory core needle biopsy of a lesion before commencing their next line of therapy. 40mL of blood will also be collected from each patient.

The biopsy sample will be run on the Pear Bio test while the patient receives their standard of care treatment. As such, for this study, the result from the Pear Bio test will not be used to inform the choice of treatment and the treating oncologist will be blinded to the test results.

The investigators will measure objective response rate (ORR) and other outcome metrics (PFS, DoR, OS, etc.). The Pear Bio test results will be compared to the actual patient outcomes to determine the test's sensitivity, specificity, positive predictive value and negative predictive value.

ELIGIBILITY:
Inclusion:

1. Able to give written informed consent prior to admission to this study.
2. Female or male aged ≥18 years.
3. Evidence of advanced RCC with intention to receive systemic therapy, defined as:

   * Clinical suspicion of advanced RCC with intention to undergo a clinically-mandated biopsy and subsequent systemic therapy OR
   * Histological evidence of advanced RCC with intention to undergo subsequent systemic therapy and willing to undergo additional research biopsy
4. At least one lesion evaluable under RECIST 1.1 criteria
5. Willing to donate at least two additional core biopsy samples prior to starting subsequent systemic therapy.
6. Willing to undergo venous sampling for 40mL of blood

Exclusion:

1. Early stage kidney cancer
2. Patients who do not have kidney cancer
3. Patients with RCC that do not intend to receive systemic therapy
4. Patients who have already commenced systemic therapy with no plans of changing the systemic therapy after the collection of the core needle biopsy.
5. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.
6. Previous diagnosis of other cancer. Previously treated cancer may be acceptable in some circumstances (e.g. surgery for an unrelated cancer > 5 years ago) after discussion with the Sponsor.
7. No lesions are amenable to biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced or metastatic kidney cancer, due to start a new line of therapy
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate correlation accuracy (sensitivity & specificity) | 6 months
  The sensitivity, specificity PPV and NPV of Pear image-based biomarkers are established against patient ORR (evaluated on imaging).

SECONDARY OUTCOMES:
Complete Response rate correlation accuracy (sensitivity & specificity) | 2 years
  The sensitivity, specificity PPV and NPV of Pear image-based biomarkers are established against patients achieving a complete response (evaluated by imaging).
Deep Response rate correlation accuracy (sensitivity & specificity) | 2 years
  The sensitivity, specificity PPV and NPV of Pear image-based biomarkers are established against patients achieving a deep response (evaluated by imaging).
Durable Response rate correlation accuracy (sensitivity & specificity) | 2 years
  The sensitivity, specificity PPV and NPV of Pear image-based biomarkers are established against patients achieving a durable response at 6, 12 and 24 months (evaluated by imaging).
PFS prediction accuracy | 2 years
  The performance of Pear image-based biomarkers are established against patients progression-free survival at 6, 12 and 24 months (evaluated by imaging).

OTHER OUTCOMES:
Culture success rate | 4 days
  The percentage of patient samples successfully arriving at central lab with >100k live cells isolated and maintaining 70% cell viability after 4 days in culture with no treatment
Hazard ratio by biomarker group | 2 years
  The hazard ratio for PFS and OS between Pear-assay biomarker-high and biomarker-low groups
OS prediction accuracy | 2 years
  The performance of Pear image-based biomarkers are established against patients overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterini Boleti, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Mount Vernon Cancer Centre, London
  - Imperial College Healthcare NHS Trust, London
  - Royal Free NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
Pseudonymised data will be shared between study sites, such as treatment and outcome data for each patient. No publication will be made revealing individual patient data; only group-level data will be published.

REFERENCES:
- Available data/document: Study Protocol — https://www.pearbio.com/peartree2

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT06264479/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT06264479/ICF_001.pdf